CLINICAL TRIAL: NCT01053468
Title: Facilitating Physical Activity Behavior and Health Outcomes in Breast Cancer Patients Receiving Chemotherapy
Acronym: PROACTIVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Athabasca University (Other)
Collaborators: University of Alberta (Other); University of Calgary (Other); Alberta Health services (Other)
Responsible Party: Jeff Vallance, PhD, Athabasca University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROACTIVE
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; physical activity; quality of life; theory of planned behavior; behavior change; health promotion
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA Behavior Intervention (Experimental): Physical Activity Resource Kit
  Interventions: Behavioral: Physical Activity Resource Kit
- Standard Materials (Active Comparator): Receive physical activity handout from the Canadian Public Health Agency
  Interventions: Behavioral: Standard Materials

INTERVENTIONS:
Behavioral: Physical Activity Resource Kit — The Intervention group (INT) will receive a Physical Activity Resource Kit which includes a step pedometer, a breast cancer-specific Physical Activity Guidebook (Exercise for health), a step pedometer resource (Step into survivorship), and a physical activity and step journal to record their daily step totals and daily physical activities.
  Participants will be instructed to wear their pedometer for the entire duration of the study (i.e., chemotherapy duration).
  Arms: PA Behavior Intervention
Behavioral: Standard Materials — Participants in this usual care group will receive a generic physical activity leaflet from the Canadian Public Health Agency
  Arms: Standard Materials

SUMMARY:
Breast cancer and its treatments can take a toll on the physical and psychosocial well-being of cancer survivors. Few interventions can help breast cancer patients improve their physical strength, stamina, and overall well-being. Developing ways to facilitate PA behavior during chemotherapy for breast cancer are necessary. This trial explores ways that breast cancer patients receiving chemotherapy can learn about and engage in PA during chemotherapy. This trial will also give Southern Alberta breast cancer survivors an opportunity to participate in evidence-based programs designed to facilitate their health, breast cancer recovery, and disease-free survival.

The investigators primary hypothesis is that women receiving the PA intervention resource kit will report a more positive change in self-reported PA at the end of chemotherapy treatments when compared to the group receiving standard materials.

DETAILED DESCRIPTION:
Primary Objective:

To compare the effects of an evidence-based intervention consisting of targeted breast-cancer specific PA print materials (i.e., Exercise for health), a step pedometer, a step-walking guidebook (i.e., Step into survivorship), and a physical activity and step journal (INT) to a comparison group receiving a generic, two-page public health PA resource (Standard Material: SM).

ELIGIBILITY:
Inclusion Criteria:

* are diagnosed with stage I -IIIA breast cancer
* are scheduled to receive neoadjuvant or adjuvant chemotherapy
* did not receive transabdominal rectus abdominus muscle (TRAM) reconstructive surgery
* are >18 years of age
* receive approval from their treating oncologist to participate
* do not have uncontrolled hypertension, cardiac illness, or psychiatric conditions (i.e., indicated in patient medical charts).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Self-reported physical activity | Baseline, post intervention, 6 months follow up

SECONDARY OUTCOMES:
Cancer specific health related quality of life | Baseline, post intervention, 6 months follow up
Psychosocial health outcomes | Baseline, post intervention, 6 months follow up
Objective step counts (pedometer) | Baseline, post intervention, 6 months follow up
Chemotherapy completion rate | Baseline, post intervention, 6 months follow up
Determinants of physical activity | Baseline, post intervention, 6 months follow up
Physical functioning | Baseline, post intervention, 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Vallance, PhD, Principal Investigator — Athabasca University
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Grande Prairie Cancer Centre, Grande Prairie, Alberta
  - Lethbridge Cancer Centre, Lethbridge, Alberta
  - Medicine Hat Cancer Centre, Medicine Hat, Alberta
  - Central Alberta Cancer Centre, Red Deer, Alberta